CLINICAL TRIAL: NCT00105209
Title: A Double-Blind, Placebo-Controlled, Three Treatment Cross-Over Study of Aspirin and Clopidogrel in Patients With Idiopathic Pulmonary Arterial Hypertension
Brief Title: A Study of Aspirin and Clopidogrel in Patients With Idiopathic Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kawut, Steven, MD (Individual)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Columbia University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HL67771-01; RR00645; RR00095; RR15534
Record Dates: First submitted 2005-03-09; First posted 2005-03-10 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Platelets
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Aspirin; Clopidogrel

INTERVENTIONS:
Drug: Aspirin
Drug: clopidogrel

SUMMARY:
Rationale: Idiopathic pulmonary arterial hypertension (IPAH) is characterized by in situ thrombosis and increased thromboxane A2 (Tx-M) synthesis. While both may be attributable to abnormal platelet function, there are no studies of anti-platelet therapy in IPAH.

Objectives: The purpose of this study is to assess the effects of aspirin (ASA) and clopidogrel on platelet function and eicosanoid metabolism in patients with IPAH.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled crossover study of aspirin 81 mg once daily and clopidogrel 75 mg once daily. Platelet function is assessed with plasma P-selectin levels and aggregometry after exposure to adenosine diphosphate, arachidonic acid, and collagen. We will assess serum levels of thromboxane B2 and urinary metabolites of thromboxane A2 and prostaglandin I2 (Tx-M and PGI-M, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPAH
* ≥ 18 years of age
* NYHA functional class I, II, or III
* Clinical stability (i.e., without change in pulmonary arterial hypertension medical regimen within one month prior to enrollment).

Exclusion Criteria:

* Other forms of PAH
* A contraindication to ASA or clopidogrel
* Thrombocytopenia (defined as platelet count ≤ 75,000)
* History of intracranial hemorrhage or chronic thromboembolic disease
* Renal failure
* Inability or unwillingness to avoid non-steroidal anti-inflammatory agents, ASA, or warfarin use for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-04; Study Completion 2003-12

PRIMARY OUTCOMES:
Plasma P-selectin level
Aggregometry
Serum thromboxane B2
Urinary Tx-M
Urinary prostaglandin I2 (PGI-M)

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia University College of Physicians and Surgeons, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee